CLINICAL TRIAL: NCT02253082
Title: Effects of OctaplasLG® on Endothelial Integrity in Patients Undergoing Emergency Surgery for Thoracic Aortic Dissections - a Randomized, Controlled, Single-blinded Investigator-initiated Pilot Trial
Brief Title: Vasculopathic Injury and Plasma as Endothelial Rescue - OCTAplas Trial (EudraCT no. 2014-000452-28)
Acronym: VIPER-OCTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Principal Investigator, Jakob Stensballe, MD, PhD, MD, PhD, Consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: VIPER-OCTA; H-3-2014-018 (Other: Regional Health Research Ethics Committee)
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Aneurysm, Thoracic; Endothelial Dysfunction
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OctaplasLG® (Active Comparator): replacement to bleeding
  Interventions: Drug: OctaplasLG®
- Standard fresh frozen plasma (Placebo Comparator): replacement to bleeding
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Drug: OctaplasLG® — OctaplasLG® is an industrial donor plasma product pooled from approximately 400 single donor units. It possess' unique features when compared to standard FFP, such as having standardized concentrations of natural pro- and anti-coagulation factors, standardized volume and as being pathogen free. Very importantly, the manufacturing method of OctaplasLG® removes immune complexes and cells in several steps of microfiltration in addition to viral, bacterial and prion pathogen inactivation.
  Other Names: Octaplas
  Arms: OctaplasLG®
Biological: Fresh frozen plasma — Standard FFP from the Blood Bank
  Other Names: FFP
  Arms: Standard fresh frozen plasma

SUMMARY:
Effects of OctaplasLG® on endothelial integrity in patients undergoing emergency surgery for thoracic aortic dissections - a randomized, controlled, single-blinded investigator-initiated pilot trial

DETAILED DESCRIPTION:
Trial Name: VIPER-OCTA trial - Vasculopathic Injury and Plasma as Endothelial Rescue - OCTAplas trial

Background

* Patients operated for thoracic aortic dissections in deep hypothermic circulatory arrest are prone to develop postoperative renal failure secondary to severe endothelial dysfunction and capillary leakage, and currently no therapy addressing this complication has proven successful
* Data from animal models of shock and massively bleeding patients indicate that plasma may be beneficial for re-establishing endothelial integrity
* Patients operated for thoracic aortic dissections generally develop requirement for massive transfusion during surgery
* Current guidelines, however, recommend against plasma transfusion to patients not needing coagulation factor replacement due to the inherent risk of transfusion complications
* OctaplasLG® is an immune complex-free and cell-free, pathogen inactivated standardized plasma product that has been shown not to be related to the transfusion complications seen secondary to standard fresh frozen plasma (FFP), thus, OctaplasLG® may be a beneficial, alternative resuscitation fluid in patients with severe endothelial dysfunction/damage
* The purpose is to bridge the knowledge gap regarding the effect of OctaplasLG® on endothelial integrity and safety

Design Single-centre randomised, single-blinded, controlled, investigator-initiated pilot trial of 42 patients undergoing emergency surgery for thoracic aortic dissections randomized to administration of OctaplasLG®, as compared to standard FFP, as coagulation factor replacement related to bleeding, when need for coagulation factor replacement is deemed necessary by the clinician according to local protocol.

Inclusion criteria

* Patient eligible for emergency surgery on cardiopulmonary bypass pump for a thoracic aortic dissections AND
* Age > 18 years AND
* Consent obtainable from patient or by proxy (independent physicians and/or next of kin)

Exclusion criteria

* Documented refusal of blood transfusion OR
* FFP transfusion before randomization OR
* Aortic dissection due to trauma OR
* Treatment with GPIIb/IIIa inhibitors < 24h from screening OR
* Withdrawal from active therapy OR
* Expected to die < 24h OR
* Previously within 30 days included in a randomized trial, if known at the time of enrolment.
* Known immunoglobulin A (IgA) deficiency with documented antibodies against IgA
* Known hypersensitivity to OctaplasLG®: the active substance, any of the excipients (Sodium citrate dihydrate, Sodium dihydrogenphosphate dihydrate or Glycine) or residues from the manufacturing process (Tri (N-Butyl) Phosphate (TNBP) and Octoxynol (Triton X-100))
* Known severe deficiencies of protein S
* Pregnancy (non-pregnancy confirmed by patient being postmenopausal or having a negative serum-hCG).

Randomization Blood Bank staff will perform 24 hour on-site randomisation by envelope-opening to allow for immediate allocation to either receiving OctaplasLG® (intervention) or standard FFP (control) as coagulation factor replacement.

Outcome measures

Primary outcome measure:

• Plasma levels of endothelial markers (Syndecan-1, soluble thrombomodulin (sTM), sE-selectin, sVE-cadherin) at 24 hours after arrival in ICU for postoperative care, as compared to baseline

Secondary outcome measures:

* Plasma levels of endothelial markers (Syndecan-1, sTM, sE-selectin, sVE-cadherin) at 48 hours postoperatively, as compared to baseline
* Acute Kidney Injury (AKI) according to RIFLE Criteria in the first 7 postoperative days, see appendix 1
* Renal replacement therapy
* Sepsis-Related Organ Failure Assessment (SOFA), worst score during ICU stay, see appendix 2
* 30-day and 90-day mortality
* P-CRP, IL-6, P-Catecholamines at 24 hours and 48 hours
* Length of stay in ICU and hospital
* Severe adverse reactions

Tertiary outcome measures

* TRALI
* TACO

Trial size The calculation is based in part by data collected in a quality control investigation of the effect of OctaplasLG® vs. FFP. The power calculation is based on the finding of a significantly higher relative level of sTM in the FFP compared to the OctaplasLG® group (p=0.025). The relative values of sTM post-CPB: FFP group: mean 3.35 (SD 2.12); OctaplasLG® group: mean 1.70 (SD 0.49); SD across the entire group of patients: 1.574. To detect the above difference with a power of 0.90 (1-β) and alpha of 0.05 requires n=21 patients in each group. The investigators have chosen to include 42 patients, 21 evaluable patients in each randomization group in case of attrition, in the present trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for emergency surgery on cardiopulmonary bypass pump for a thoracic aortic dissections AND
* Age > 18 years AND
* Consent obtainable from patient or by proxy (independent physicians and/or next of kin)

Exclusion Criteria:

* Documented refusal of blood transfusion OR
* FFP transfusion before randomization OR
* Aortic dissection due to trauma OR
* Treatment with GPIIb/IIIa inhibitors < 24h from screening OR
* Withdrawal from active therapy OR
* Expected to die < 24h OR
* Previously within 30 days included in a randomized trial, if known at the time of enrolment
* Known IgA deficiency with documented antibodies against IgA
* Known hypersensitivity to OctaplasLG®: the active substance, any of the excipients (Sodium citrate dihydrate, Sodium dihydrogenphosphate dihydrate or Glycine) or residues from the manufacturing process (Tri (N-Butyl) Phosphate (TNBP) and Octoxynol (Triton X-100))
* Known severe deficiencies of protein S
* Pregnancy (non-pregnancy confirmed by patient being postmenopausal or having a negative serum-hCG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-11; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma levels of endothelial markers (Syndecan-1, sTM, sE-selectin, sVE-cadherin) | At 24 hours after arrival in ICU for postoperative care, as compared to baseline

SECONDARY OUTCOMES:
Plasma levels of endothelial markers (Syndecan-1, soluble thrombomodulin (sTM), sE-selectin, sVE-cadherin) | At 48 hours postoperatively, as compared to baseline
Acute Kidney Injury (AKI) according to RIFLE Criteria | In the first 7 postoperative days
Renal replacement therapy | In the first 7 postoperative days
Sepsis-Related Organ Failure Assessment (SOFA) | Worst score In the first 7 postoperative days
Mortality | 30-day and 90-day
P-Creactive protein (CRP), Interleukin-6 (IL-6), P-Catecholamines | At 24 hours and 48 hours
Length of stay in ICU and hospital | Days, assessed at 30-days and 90-days
Severe adverse reactions | In the first 30 postoperative days

OTHER OUTCOMES:
Transfusion associated acute lung injury (TRALI) | In the first 30 postoperative days
Transfusion associated circulatory overload (TACO) | In the first 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stensballe, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stensballe J, Ulrich AG, Nilsson JC, Henriksen HH, Olsen PS, Ostrowski SR, Johansson PI. Resuscitation of Endotheliopathy and Bleeding in Thoracic Aortic Dissections: The VIPER-OCTA Randomized Clinical Pilot Trial. Anesth Analg. 2018 Oct;127(4):920-927. doi: 10.1213/ANE.0000000000003545. PMID 29863610